CLINICAL TRIAL: NCT05479942
Title: Impact of Graded Motor Imagery Training Paradigm on Shoulder Pain and Quality of Life in Patients With Chronic Stroke
Brief Title: Graded Motor Imagery Training Paradigm on Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohammed samir (Other)
Responsible Party: Sponsor-Investigator, Mohammed samir, Assistant lecturer, Merit University
Organization: Merit University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1255
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Stroke, Complication
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Study group
  Interventions: Other: Graded motor imagery training paradigm; Other: conventional therapy (task-oriented active/passive range of motion training)
- Group B (Experimental): Control group
  Interventions: Other: conventional therapy (task-oriented active/passive range of motion training)

INTERVENTIONS:
Other: Graded motor imagery training paradigm — Graded motor imagery is the psychological representation of attention doing movement of a part of body, without actually moving that part, it broken down into three unique stages of treatment techniques:
  1. Left/right discrimination (Implicit motor imagery):
  2. Explicit motor imagery
  3. Mirror Therapy
  Arms: Group A
Other: conventional therapy (task-oriented active/passive range of motion training) — Patient will do 3 tasks as: drinking water from a glass, lifting a glass of water to a level of 90° shoulder flexion with an extended elbow, moving 5 crystals from the table to a box, wiping the table with a towel with the elbow extended, grasping and releasing a 6 cm in diameter tennis ball, and combing their hairs.
  Practice shoulder flexion and abduction active ROM, and passive ROM training

SUMMARY:
Background: Shoulder pain is the most common pain disorder after stroke and one of the most common complications reduced quality of life. Graded Motor Imagery (GMI) is the most up to date rehabilitation program - based on the latest science and clinical trials - to treat many complex pain, and movement problems. Graded motor imagery is the psychological representation of attention doing movement of a part of body, without actually moving that part, it broken down into three unique stages of treatment techniques:

1. Left/right discrimination: The ability to identify left or right images of their painful body parts. This ability appears to be important for normal recovery from pain. The good news is that the brain is plastic and changeable, if given the right training for long enough.
2. Explicit motor imagery: Essentially thinking about moving without actually moving. Imagined movements can actually be hard work if in pain. This is most likely because 25 percent of the neurons in brain are 'mirror neurons' and start firing when thinking of moving or even watch someone else move. By imagining movements, use similar brain areas as actually move. This is why sports people imagine an activity before they do it.
3. Mirror therapy: If putting person left hand behind a mirror and right hand in front, person can trick brain into believing that the reflection of right hand in the mirror is left. Person is now exercising left hand in the brain, particularly if person start to move right hand. Graded motor imagery training has been suggested as a treatment technique that should be utilized in addressing shoulder pain and movement impairments following stroke.

DETAILED DESCRIPTION:
Stroke is one of the main causes of mortality and disability in the world, and it was reported that about 15 million people suffer from stroke each year, which impose a heavy burden on social health care system. Meanwhile, shoulder pain after stroke, a common and disabling complication, with a prevalence of up to 12%-49%. Usually occurs two to three months after stroke and may result in withdrawal from rehabilitation programs, longer hospital stays, reduced limb function, impairing quality of life of the stroke patients adversely.

Stroke patients with poor upper extremity function have an increased risk of hemiplegic shoulder pain. Various theories have been proposed for the development of hemiplegic shoulder pain, including deficiency in pain adaption , central sensitization to normal or sub-threshold sensory stimuli, and impaired neuromuscular control of the scapula.

Graded motor imagery process from innovation of improved sensory cortex organization to targeted sensory discrimination exercise for clinical benefit has been frequent in complex regional pain syndrome (CRPS). Without eliciting the protective response of pain graded motor imagery slowly involves cortical motor networks. Excessively complex nociception system and the interrupted cortical mechanisms are only provided by graded motor imagery.

Graded motor imager (GMI) uses have 3 sequential stages for application. Left and right judgment which activates premotor cortex without activating primary motor areas is the first stage of graded motor imagery. Fictional movements which trigger motor cortical parts similar to those activated in actual accomplishment of movement is the second stage of graded motor imagery. Mirror therapy triggers not only motor cortex but also provides a strong visual input to the cortex in the third or final stage of graded motor imagery, though activation for each stage of GMI have been supported by brain imaging in healthy subjects.

Statement of the problem:

This study will try to answer the following question:

Will Graded motor imagery training paradigm be effective in the treatment of shoulder pain?

Purpose of the study:

The purpose of this study was designed to investigate the effect of graded motor imagery training paradigm in treatment shoulder pain and quality of life.

Significant of the study:

Shoulder pain is the most common pain disorder after stroke and one of the four most common complications. The estimated incidence ranges from of 30-70%. Shoulder pain is associated with reductions in function, interference with rehabilitation efforts, and a reduced quality of life.

Onset of shoulder pain is rapid, occurring as soon as a week after stroke in 17% of patients. While shoulder pain is ubiquitous, the management of shoulder pain represents a complex treatment pathway with insufficient evidence supporting one particular treatment .

Multiple factors contribute to normal shoulder positioning and function. Proper shoulder positioning involves a stabilized glenohumeral joint (actively and passively), appropriate glenoid fossa angle, and correct scapular and vertebral column alignment. The suprascapular nerve is not only vital to motor function, it provides up to 70% of the sensory fibers to the shoulder, and pain transmitted by the suprascapular nerve represents another potential underlying cause of shoulder pain.

Graded motor imagery it is very good method in pain management that organizes cortical activation and gradually decreases cortical disinhibition to prevent from acute pain to chronic pain.A non-randomized trial demonstrated some effect of GMI on motor function in patients with chronic stroke.

GMI has been extensively studied in chronic pain patients, especially chronic regional pain syndrome (CRPS) .It was developed to grade cortical activa¬tion and to reduce cortical disinhibition in CRPS. Cortical disinhibition is surely one of the patho-physio¬logical consequences of stroke that contributes to motor impairment. Stroke and CRPS have been compared on other grounds too.GMI has been suggested as a treatment technique that should be utilized in address¬ing movement impairments following stroke.

Graded motor imagery is the psychological representation of attention doing movement of a part of body, without actually moving that part. Because of this, it was intended to conclude the effects of graded motor imagery (GMI) training paradigm on shoulder pain and disability in chronic stroke patients.

Delimitations:

Patients were delimited to:

1. Forty two patients who had chronic Stroke.
2. Age ranged from 45 to 65 years old males and females.
3. The patients were randomly divided into two groups of equal number.
4. Patients have shoulder pain and functional disability due to chronic stroke.
5. Patients will be assessed via Recognise Online program for speed and accuracy of responses, Shoulder Pain and Disability Index (SPADI) for pain and function, and electrical goniometer for shoulder Range of Motion (ROM).
6. Patients will receive Graded motor imagery training paradigm and conventional therapy (task-oriented active/passive range of motion training).

Basic Assumption:

It was assumed that:

1. All patients followed the instructions that were given to them.
2. The measurement tools were reliable and valid.
3. All patients were free from cognitive or psychological disorders.
4. All patients were free from any systemic disease or its complication that affects the therapeutic out.

Hypothesis:

There was no effect of Graded motor imagery on shoulder pain and quality of life in patients with chronic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 45 to 65 years old.
2. All patients suffer from shoulder pain post chronic stroke.
3. All patients received same kind of medications.
4. All patients have shoulder mild subluxation diagnosed by X- ray

4. All patients with modified Ashworth scale up to grade 2 muscle tone.

Exclusion Criteria:

1. Patient who suffers from shoulder stiffness post chronic stroke.
2. Patient who suffers from bilateral shoulder pain due to multiple stroke.
3. Patient who suffers from loss of hand movement post stroke.
4. Patient who suffers from mental or psychological disorders.
5. Patient dropped out through the study more than three sessions.
6. Patient who suffers from any systemic disease that may interfere with the objectives of the study

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Recognise Online program | up to 8 weeks
  The Recognise online application that displays different parts of the body that correspond to the patients' affected limb (left, right). During this portion of GMI, a patient is shown a group of images that correspond to the affected limb.four values for speed and four for the accuracy of responses corresponding to each patient for each treatment session
Flexible electronic goniometer | up to 8 weeks
  To assess shoulder range of motion, while the patient was sitting down on a chair. The measurement involved the active flexion and abduction of the shoulder, with the upper limb starting from the neutral position.In each session, there were two measurements, The first was done at the beginning of the session and the second at the end of the session
The Shoulder Pain and Disability Index (SPADI) | up to 8 weeks
  It is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder every session

CONTACTS AND LOCATIONS:
Overall Officials: Nawal Abo Shady, professor, Study Director — Professor of Physical Therapy Cairo University
Locations (1):
- El Baliana Central Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be available for improve clinical research
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication after july 2024 for ever
Access Criteria: free for all